CLINICAL TRIAL: NCT04759911
Title: Neoadjuvant Treatment With Selpercatinib in RET-Altered Thyroid Cancers
Brief Title: Selpercatinib Before Surgery for the Treatment of RET-Altered Thyroid Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0570; NCI-2021-00535 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0570 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-02-08; First posted 2021-02-18 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Malignant Thyroid Gland Neoplasm; Poorly Differentiated Thyroid Gland Carcinoma; Recurrent Thyroid Gland Carcinoma; Thyroid Gland Anaplastic Carcinoma; Thyroid Gland Medullary Carcinoma; Thyroid Gland Papillary Carcinoma; Thyroid Gland Squamous Cell Carcinoma
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Carcinoma, Anaplastic; Carcinoma, Medullary; Thyroid Cancer, Papillary | interventions — selpercatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (selpercatinib) (Experimental): Patients receive selpercatinb PO BID on days 1-28. Treatment repeats every 28 days for up to 7 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care surgery.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Selpercatinib; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Selpercatinib — Given PO
  Other Names: LOXO-292; RET Kinase Inhibitor LOXO-292; Retevmo; WHO 10967
Procedure: Therapeutic Conventional Surgery — Undergo standard of care surgery

SUMMARY:
This phase II trial studies the effect of selpercatinib given before surgery in treating patients with thyroid cancer whose tumors have RET alterations (changes in the genetic material [deoxyribonucleic acid (DNA)]). Selpercatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving selpercatinib before surgery may help shrink the tumors and help control the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the efficacy of neoadjuvant selpercatinib in medullary thyroid cancer by objective response rate (ORR) per RECIST (standard Response Evaluation Criteria in Solid Tumors [RECIST]).

SECONDARY OBJECTIVES:

I. To evaluate the efficacy of neoadjuvant selpercatinib in medullary thyroid cancer by ORR per modified neck RECIST.

II. To evaluate the efficacy of neoadjuvant selpercatinib in medullary thyroid cancer per surgical margin status, which is categorized as R0, R1, and R2 surgical resection.

III. To evaluate the safety profile of neoadjuvant selpercatinib.

IV. To evaluate the efficacy of neoadjuvant selpercatinib on progression-free survival (PFS), including overall PFS and locoregional PFS.

V. To measure changes in expected and actual surgical morbidity/complexity as well as evaluate changes of R0/R1 resection rates in pre-specified extrathyroidal anatomic target interfaces before and after selpercatinib treatment.

EXPLORATORY OBJECTIVES:

I. In patients with differentiated thyroid cancer [DTC] and anaplastic thyroid cancer [ATC] only, to evaluate the efficacy of neoadjuvant selpercatinib by ORR per RECIST (standard RECIST and modified neck RECIST), surgical margin status (R0/R1 versus [vs.] R2), safety profile, surgical morbidity/complexity, PFS and overall survival (overall survival [OS], ATC only).

II. To define and measure changes of patient-reported outcomes and quality of life as measured by MD Anderson Symptom Inventory (MDASI) and European Quality of Life Five Dimension (EQ-5D) in patients with RET-altered thyroid cancer who receive selpercatinib treatment.

III. To explore translational endpoints in selpercatinib neoadjuvant therapy with biopsies/tissue collection before selpercatinib treatment and during surgery.

IV. To explore peripheral and tissue measures associated with selpercatinib mechanisms of resistance in patients who experience disease progression after selpercatinib treatment.

OUTLINE:

Patients receive selpercatinb orally (PO) twice daily (BID) on days 1-28. Treatment repeats every 28 days for up to 7 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care surgery.

After completion of study treatment, patients are followed up for disease progression status every 3-4 months for the first 2 years. ATC patients continue follow-up every 6 months for year 3 and 4, and once in year 5.

ELIGIBILITY:
Inclusion Criteria:

* Patients with RET-altered thyroid cancer who present with locally advanced primary tumor, defined as T3 or T4 by imaging or invasive/bulky nodal disease, or with recurrent/residual invasive/bulky nodal disease will be enrolled in this trial, regardless of whether distant metastases are present or not
* At least 12 years of age on the day of signing informed consent
* Pathologic findings supporting the clinical impression of medullary thyroid carcinoma, papillary thyroid carcinoma, poorly differentiated thyroid carcinoma, or anaplastic thyroid carcinoma. Diagnosis of anaplastic thyroid carcinoma may include consistent with or suggestive of terminology associated with: anaplastic thyroid carcinoma, undifferentiated carcinoma, squamous carcinoma; carcinoma with spindled, giant cell, or epithelial features; poorly differentiated carcinoma with pleomorphism, extensive necrosis with tumor cells present
* Having an activating RET gene alteration (fusion or mutation). The RET alteration result should be generated from a laboratory with Clinical Laboratory Improvement Act (CLIA), ISO/EIC, College of American Pathologists (CAP), or other similar certification that clearly denotes the presence of a RET alteration in tumor, or institutional-approved cell free DNA blood test for RET alteration
* Prior multikinase inhibitors (MKIs) with anti-RET activity are allowed. The specific agent(s), duration of treatment, clinical benefit, and reason for discontinuation (e.g., progressive disease [PD], drug toxicity, or intolerance) should be documented for all kinase inhibitors the patient has been exposed to
* At least one measurable lesion as defined by RECIST 1.1
* Surgical morbidity/complexity score of 1 to 4 (moderate, severe, very severe, or unresectable)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 (age >= 16 years) or Lansky Performance Score (LPS) >= 40% (age < 16 years) with no sudden deterioration 2 weeks prior to study registration
* Absolute neutrophil count (ANC) >= 1500/uL
* Hemoglobin >= 9 g/dL (5.58 mmol/L)
* Platelets >= 100,000/uL
* Total bilirubin =< 1.5 X upper limit of normal (ULN) (Except participants with a documented history of Gilbert syndrome who must have a total bilirubin < 3 X ULN)
* Alanine Aminotransferase (ALT)/Aspartate Aminotransferase (AST) < 2.5 X ULN OR < 5 X ULN if the liver has tumor involvement
* Normal serum potassium, calcium, and magnesium levels (may be receiving supplements). Grade 1 hypocalcemia (corrected serum calcium > 8) is acceptable
* Willing to undergo tumor biopsy prior to trial treatment, unless in the opinion of the treating physician, a biopsy is not feasible or safe. Subjects must be willing to ultimately undergo surgery if their tumor becomes surgically resectable
* Ability to comply with outpatient treatment, laboratory monitoring, and required clinic visits for the duration of study participation
* Willing and able to provide written informed consent signed by study patient (or legally acceptable representative if applicable)
* Willingness of men with partners of childbearing potential or women of childbearing potential to use a highly effective contraceptive method during treatment with study drug and for 3 months following the last dose of study drug. Male study participants should refrain from sperm donation during study treatment and for up to 6 months following the last dose of selpercatinib

Note:

* Unless not allowed by local regulations, women of childbearing potential who are abstinent (if this is complete abstinence, as their preferred and usual lifestyle) or in a same-sex relationship (as part of their preferred and usual lifestyle) must agree to either remain abstinent or stay in a same-sex relationship without sexual relations with males. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post ovulation methods), declaration of abstinence just for the duration of the trial, and withdrawal are not acceptable methods of contraception
* A postmenopausal woman will be defined as having no menses for 12 months without an alternative medical cause. Male sterility will be defined as only men sterilized surgically. For male patients with a pregnant partner, a condom should be used for contraception. For male patients with a non-pregnant female partner of child-bearing potential and woman of childbearing potential one of the following birth control methods with a failure rate of less than 1% per year when used consistently and correctly are recommended:

  * Combined estrogen and progesterone containing hormonal contraception associated with inhibition of ovulation given orally, intravaginally, or transdermally
  * Progesterone-only hormonal contraception associated with inhibition of ovulation given orally, by injection, or by implant
  * Intrauterine device (IUD)
  * Intrauterine hormone-releasing system (IUS)
  * Bilateral tubal occlusion
  * Vasectomized partner
  * Sexual abstinence

    * Women of childbearing potential must have a negative pregnancy test (serum) documented at screening and then negative serum or urine pregnancy testing at day 1 of every treatment cycle (exception: negative pregnancy testing within 21 days prior to cycle 1 day 1 [C1D1] is allowed)

Exclusion Criteria:

* An additional validated oncogenic driver that could cause resistance to selpercatinib treatment (if known)
* Prior treatment with a selective RET inhibitor(s) (pralsetinib [BLU-667], including investigational selective RET inhibitor[s])
* Investigational agent or anticancer therapy (including chemotherapy, biologic therapy, or immunotherapy) within 5 half-lives or 3 weeks (whichever is shorter) prior to planned start of selpercatinib

  * Exception: Patients with ATC
* No concurrent investigational anti-cancer therapy is permitted
* Major surgery (excluding placement of vascular access and diagnostic procedures) within 4 weeks prior to planned start of selpercatinib

  * Exception: Patients with ATC
* Radiotherapy with a limited field of radiation for palliation within 1 week of the first dose of study treatment, with the exception of patients receiving radiation to more than 30% of the bone marrow or with a wide field of radiation, which must be completed at least 4 weeks prior to the first dose of study treatment
* Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of starting study treatment with the exception of alopecia and grade 2, prior platinum therapy related neuropathy
* Symptomatic primary central nervous system (CNS) tumor, metastases, leptomeningeal carcinomatosis, or untreated spinal cord compression

  * Exception: Patients are eligible if neurological symptoms and CNS imaging are stable and steroid dose is stable for 14 days prior to the first dose of selpercatinib and no CNS surgery or radiation has been performed for 28 days, 14 days if stereotactic radiosurgery (SRS)
* Patients with clinically significant active cardiovascular disease, Torsades de pointes, or history of myocardial infarction within 6 months prior to planned start of study treatment or prolongation of the QT interval corrected for heart rate using Fridericia's formula (QTcF) > 470 msec
* Patients with clinically significant active malabsorption syndrome or other condition likely to affect gastrointestinal absorption of the drug
* Use of a concomitant medication that is known to cause QTc prolongation
* Active uncontrolled systemic bacterial, viral, or fungal infection, or serious ongoing intercurrent illness, such as uncontrolled hypertension (systolic blood pressure [BP] >= 140 mmHg or diastolic BP >= 90 mmHg per CTCAE) or diabetes, despite optimal treatment. Screening for chronic conditions is not required
* Uncontrolled symptomatic hyperthyroidism or hypothyroidism

  * Exception: Patients with papillary thyroid cancer (PTC)
* Uncontrolled symptomatic hypercalcemia or hypocalcemia
* Pregnancy or lactation
* Active second malignancy other than minor treatment of indolent cancers

  * Exception: Patients with PTC or patients with stable pheochromocytoma in MEN2
* History of severe hypersensitivity (>= grade 3) to selpercatinib and/or any of its excipients

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-02-26 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 7 months
  Defined as the percentage of number of complete response or partial response in total number of patients treated. With ORR by Response Evaluation Criteria in Solid Tumors (RECIST), will report the percentages of patients that fall into each of the four categories: complete response, partial response, stable disease or progressive disease according to RECIST 1.1.
Tumor response | Up to 7 months
  Assessed using modified neck RECIST, which applies the RECIST criteria only to lesions above the clavicles. Will report the percentages of patients that fall into each of the four categories: complete response, partial response, stable disease or progressive disease according to modified neck RECIST 1.1.

SECONDARY OUTCOMES:
R0/R1 resection rates | During surgery
  Defined by proportion of patients who undergo successful thyroidectomy with clear (R0) or microscopically positive (R1) surgical margins. Will evaluate R0/R1 resection rates in each of 4 pre-specified extrathyroidal anatomic target interfaces: 1) perithyroid muscles (e.g. strap, sternocleidomastoid, inferior constrictor muscles) 2) cartilage (larynx/trachea) 3) esophagus 4) recurrent laryngeal nerve.
Progression free survival (PFS) | Up to 2 years post treatment
  Defined as the time from patient registration to disease progression or death from any cause. Structural progression is defined according to RECIST criteria based on histopathologic findings, and biochemical progression is defined as abnormal thyroglobulin (Tg) or rising Tg antibody levels for anaplastic thyroid cancer/differentiated thyroid cancer, and abnormal carcinoembryonic antigen/calcitonin for medullary thyroid cancer.
Locoregional PFS | Up to 2 years post treatment
  Defined as the time from patient registration to locoregional progression or death from any cause. Locoregional progression is defined as disease progression above the clavicles according to modified neck RECIST criteria.
Surgical morbidity/complexity score | Baseline to the date of surgery, assessed up to 7 months
  Surgical morbidity/complexity score will be measured at enrollment, prior to surgery and at surgery. The Thyroid Neck Group Morbidity Complexity Scoring and MGH/MEE-MSK-MD Anderson (MMM) Surgical Morbidity Complexity Score are incorporated, specifying on scale with 5 levels of complexity and mobidity of the surgery [mild (level 0), moderate (level 1), severe (level 2), very severe (level 3), and unresectable (level 4)]. The surgical morbidity/complexity scores will be collected at enrollment, prior to surgery and at surgery; descriptive statistics such as means and standard deviations will be calculated for each time point.
Overall survival (OS) | Up to 5 years post treatment
  Defined as the time from patient registration to death from any causes.
Incidence of adverse events | Up to 7 months
  Assessed as defined by Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0.
Quality of life | Up to 2 years post treatment
  Assessed by the European Quality of Life 5 Dimension Questionnaire (EQ-5D). The EQ-5D consists of health state description and evaluation. The health state description consists of five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), with each dimension specifying five levels of severity [best (1)-worst (5)]. The health state evaluation is assessed using the visual analogue scale ([worse (0)-best (100)].
Patient-reported outcomes | Up to 2 years post treatment
  Measured by the M.D. Anderson Symptom Inventory for Head and Neck Cancer (MDASI-HN) instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Zafereo, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - University of Michigan Health Systems, Ann Arbor, Michigan
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org